CLINICAL TRIAL: NCT02763631
Title: Symptomatic Treatment of Excessive Dynamic Airway Collapse Using Daytime Portable Continuous Positive Airway Pressure
Acronym: EPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: B&D Electromedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/LO/0028
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Excessive Dynamic Airway Collapse; Tracheobronchomalacia
MeSH Terms: conditions — Tracheobronchomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Run In Phase (Experimental): Eligible patients will have 6-Minute Walk Test (6-MWT) on self ventilation and on CPAP
  Interventions: Other: Experimental: Run In Phase
- Treatment (Experimental): Those patients who improve their 6-MWT by more than 30 meters will then be randomised to either:
  Treatment arm - Patients will be setup onto portable CPAP during the day
  Interventions: Other: Experimental: Treatment
- Standard Care Arm (Sham Comparator): Those patients who improve their 6-MWT by more than 30 meters will then be randomised to either:
  Control Arm - Standard care arm.
  Interventions: Other: Sham Comparator: Stand Care Arm

INTERVENTIONS:
Other: Experimental: Treatment — Participants will be established on portable CPAP during the day with nasal pillows as an interface and requested to use it at least 8 hours/day.
  Arms: Treatment
Other: Experimental: Run In Phase — Participants will undergo a run-in phase during which they will undergo baseline assessments. If they tolerate the portable CPAP and if their 6-MWT improves by more than 30m when performed on CPAP, they will be randomised into the trial.
  Arms: Run In Phase
Other: Sham Comparator: Stand Care Arm — No change will be made to participants care
  Arms: Standard Care Arm

SUMMARY:
The aim of this study is to assess the benefit of a portable ventilator generating positive end-expiratory pressure on exercise tolerance in patients with Excessive dynamic airway collapse (EDAC) and tracheobronchomalacia (TBM).

DETAILED DESCRIPTION:
Excessive dynamic airway collapse (EDAC) and tracheobronchomalacia (TBM) occur due to abnormal weakening of the walls of the central airways leading to central airway collapse on expiration. This collapse is responsible for breathlessness, cough or syncope. In adults, this weakening can be idiopathic (Mounier-Khun syndrome), secondary to respiratory diseases such as chronic obstructive pulmonary disease (COPD), secondary to systemic diseases such as relapsing polychondritis (RP) or secondary to invasive ventilation or trauma. The incidence of EDAC and TBM varies from 12% in all patients undergoing bronchoscopy to 44% in patients with chronic bronchitis undergoing bronchoscopy. Gold standard for the diagnosis of EDAC and TBM is bronchoscopy which identifies and quantifies the narrowing of the airway. Non-invasive technique such as inspiratory and expiratory chest computed-tomography (CT) can also be used to diagnose EDAC / TBM.

Currently, in addition to management of the underlying disease, treatment options for EDAC / TBM are limited. Surgical tracheoplasty can be offered but can be associated with severe post-operative complications. Airway stenting can also be offered but, even if this treatment improved quality of life, it fails to improve exercise capacity. Airway stenting is also associated with infectious complications as well as stent migrations. Other endoscopic treatment such as Yttrium Aluminium Perovskite laser can be offered with good results but have not yet been validated in a randomised trial. Nocturnal non-invasive ventilation (NIV) can also be used, especially in patients with associated obstructive sleep apnoeas but again there is not randomised clinical trial evidence that validates this approach in adults. Expiratory Positive Airway Pressure (EPAP) provides a pneumatic stenting that prevents the expiratory collapse of the airway. But, by giving the NIV during the night, patients are left without any support during the day whilst their respiratory demand is higher and when they are more symptomatic. Currently, NIV is only given at night or at rest because current non-invasive ventilators are not suitable for ambulatory use as they are heavy. Recently, a new portable ventilator with built-in battery has been issued (Z1®, Breas®). This ventilator is light (500g) portable and has a working duration of 8 hours. Therefore, it can be easily carried and used while walking. By providing a nasal pillow interface (Nasal swift®, Resmed®) to patients, it will allow them to walk safely with the device on.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed EDAC or TBM on inspiratory/expiratory CT or bronchoscopy
* Patient with exertional dyspnea

Exclusion Criteria:

* Pregnancy
* Significant physical or psychiatric comorbidity that would prevent compliance with trial protocol
* Inability to perform 6-MWT
* Current intra-tracheal stent
* Previous surgery for EDAC or TBM
* Uncontrolled underlying disease:

  * Initiation of home mechanical ventilation in last 3 months
  * Uncontrolled joint pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Does daytime activity by an accelerometer change from baseline to 4 weeks | 4 weeks
  Daytime activity assessed by an accelerometer. Participants will be assessed at baseline and at 4 weeks in the control arm and in the treatment arm with participants on portable CPAP to see if there is any change between the time frames and between the groups on daytime activity measured by accelerometers that all participants randomised into the trial will wear from baseline to follow up at 4 weeks.

SECONDARY OUTCOMES:
Distance in 6-MWT on Continous Positive Airway Pressure (CPAP) at 4 weeks follow-up | 4 weeks
  Is there a change in exercise capacity measured by 6-MWT for all patients in the study from baseline to 4 weeks. All walk tests will be performed on portable Continuous Positive Airway Pressure (CPAP)
Change in respiratory-related quality of life - Severe Respiratory Insufficiency (SRI) | 4 weeks
  Is there a change in quality of life from baseline to 4 weeks measured by Severe Respiratory Insufficiency Questionnaire
Change in respiratory-related quality of life - St George's Respiratory Questionnaire (SGRQ) | 4 weeks
  Is there a change in quality of life from baseline to 4 weeks measured by St George's Respiratory Questionnaire.
Change in neural respiratory drive with parasternal electromyography | 4 weeks
  Is there a change in neural respiratory drive measured by parasternal electromyography both at rest and whilst using portable CPAP at baseline and at 4 weeks
Change of lung homogeneity assessed by electrical impedance tomography while on CPAP | 4 weeks
  Is there a change in lung homogeneity in participants from baseline to 4 weeks. Measured by electrical impedence tomography whilst all participants are using portable CPAP
Change in cross-sectional area quadriceps rectus femoris ultra-sound | 4 weeks
  Is there a change in the area of the quadriceps rectus femoris in participants from baseline to 4 weeks. Measured using ultrasound which will be performed on all participants

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No